CLINICAL TRIAL: NCT02462668
Title: The Efficiency and Safety of Fibreoptic Bronchoscopy Assisted Intubation During Noninvasive Positive Pressure Ventilation
Brief Title: Fibreoptic Bronchoscopy Assisted Intubation During Noninvasive Positive Pressure Ventilation
Acronym: FBAIDNIPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lingbo Nong (Other)
Responsible Party: Sponsor-Investigator, Lingbo Nong, MD, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LNong
Record Dates: First submitted 2015-05-24; First posted 2015-06-04 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Respiratory Failure
Keywords: Bronchoscopy; Intubation; Noninvasive positive pressure ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Preoxygenation with Bag-mask ventilation before fibreoptic bronchoscopy assisted intubation.
  Intervention: Bag-mask ventilation.
  Interventions: Procedure: Bag-mask ventilation; Procedure: fibreoptic bronchoscopy assisted intubation
- NIPPV (Experimental): The NIPPV group preoxygenation with noninvasive positive pressure ventilation(NIPPV), And then receives fibreoptic bronchoscopy intubation through a face mask (there is a small hole allow to insert the tracheal tube through the mask into trachea) during NIPPV.
  Intervention: noninvasive positive pressure ventilation(NIPPV)
  Interventions: Procedure: Noninvasive positive pressure ventilation(NIPPV); Procedure: fibreoptic bronchoscopy assisted intubation

INTERVENTIONS:
Procedure: Bag-mask ventilation — The control group receives preoxygenation with bag-mask ventilation
  Arms: Control
Procedure: Noninvasive positive pressure ventilation(NIPPV) — The NIPPV group receives noninvasive positive pressure ventilation during fibreoptic bronchoscopy assisted intubation
  Arms: NIPPV
Procedure: fibreoptic bronchoscopy assisted intubation — All patients will receive fibreoptic bronchoscopy assisted intubation.

SUMMARY:
This study is to investigate the efficiency and safety of fibreoptic bronchoscopy assisted intubation during noninvasive positive pressure ventilation in respiratory failure patients. Half of the participants will receive preoxygenation with noninvasive ventilator and fibreoptic bronchoscopy intubation during NIPPV. While the other half using usual preoxygenation(bag-mask ventilation ).

DETAILED DESCRIPTION:
Respiratory failure is very common for critically ill patients, Main complication associated with intubation was desaturation. Usual preoxygenation( bag-mask ventilation) have been show that marginally effective in critically ill patients. As a result, there is a need to optimize the technique of preoxygenation to prolong the safe duration of apnea during the intubation procedure in critically ill patients. Noninvasive ventilation provides continuous positive airway pressure is effective in increasing the efficiency of gas exchange and in reducing the decrease in oxyhemoglobin saturation during fiberoptic bronchoscopy in hypoxemic patients.

Therefore, our aim was to study whether NIPPV is more effective at reducing desaturation than usual preoxygenation in hypoxemic, critically ill patients requiring intubation in ICU.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure requiring intubation,
* Age greater than or equal to 18 years

Exclusion Criteria:

1. Nasal polyps，Nasopharyngeal cancer，Nasal bleeding，Rhinitis，Sinusitis and so on Nasal disease
2. Basal skull fracture
3. Severe coagulopathy, blood platelet counts <50×10*9/L
4. Nose and facial deformities, trauma
5. Cardiac arrest
6. Pregnancy or puerpera

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06-11 (Actual); Study Completion 2017-06-18 (Actual)

PRIMARY OUTCOMES:
Change in pulse oxymetry(SpO2) | From time of randomization until connect to ventilator 30min

SECONDARY OUTCOMES:
Mechanical ventilation Time | 28 days

OTHER OUTCOMES:
28 days survival rate | From the day of intubation to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, investigator, Study Director — The First Hospital Of Guangzhou Medical college
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Nong L, Liang W, Yu Y, Xi Y, Liu D, Zhang J, Zhou J, Yang C, He W, Liu X, Li Y, Chen R. Noninvasive ventilation support during fiberoptic bronchoscopy-guided nasotracheal intubation effectively prevents severe hypoxemia. J Crit Care. 2020 Apr;56:12-17. doi: 10.1016/j.jcrc.2019.10.017. Epub 2019 Nov 14. PMID 31785505